CLINICAL TRIAL: NCT06271369
Title: A Real-world Study Comparing Tisagenlecleucel (Tisa-cel) With Axicabtagene Ciloleucel (Axi-cel) on Healthcare Resource Use (HRU), Costs, and Overall Survival (OS) in Diffuse Large B-cell Lymphoma (DLBCL): A Retrospective Study of Medicare Population
Brief Title: Real-World HRU and Costs in DLBCL Pts With Tisa-cel and Axi-cel, a Medicare Study.
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CCTL019CUS13
Record Dates: First submitted 2024-02-14; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Diffuse Large B-cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Tisa-cel cohort: Patients with at least one ICD-10 diagnosis for DLBCL who were at least 18 years old. Patients also had at least three months of continuous health plan enrollment before administration of CAR-T therapy and received tisa-cel following DLBCL diagnosis.
- Axi-cel cohort: Patients with at least one ICD-10 diagnosis for DLBCL who were at least 18 years old. Patients also had at least three months of continuous health plan enrollment before administration of CAR-T therapy and received axi-cel following DLBCL diagnosis.

SUMMARY:
This was a retrospective non-interventional cohort study design using the Centers for Medicare and Medicaid Services (CMS) 100% Medicare data (2015Q1-2020Q4).

Eligible adult patients with r/r DLBCL who were treated with CAR-T therapy were identified from the CMS 100% Medicare data. Patients who received chimeric antigen receptor modified T cell (CAR-T) therapy were further classified into tisa-cel and axi-cel cohorts based on the type of CAR-T treatment received. The index date was defined as the date of tisa-cel or axi-cel therapy administration. Baseline period was defined as three months prior to the index date. Study period was defined from the index date to the end of health plan coverage based on insurance enrollment file or death, whichever occurred earlier.

ELIGIBILITY:
Inclusion Criteria:

* Patients had at least one International Classification of Diseases, 10th Revision (ICD-10) diagnosis code for DLBCL.
* Patients received CAR-T therapy, including both tisa-cel and axi-cel, following DLBCL diagnosis. The administration date of CAR-T therapy was defined as the index date.
* Patients were at least 18 years of age as of the index date.
* Patients had at least three months of continuous health plan enrollment before the index date.

Exclusion Criteria:

* Patients who had a medical claim associated with a clinical trial within one month before and after the index date.
* Patients who had zero cost on index date for CAR-T infusion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 613 (Actual)
Dates: Start 2022-08-11 (Actual); Primary Completion 2023-02-15 (Actual); Study Completion 2023-02-15 (Actual)

PRIMARY OUTCOMES:
Number of patients with IP admission | Up to approximately 6 years
Number of IP admissions | Up to approximately 6 years
IP days | Up to approximately 6 years
  Described as the cumulative number of days during IP stays including ICU.
Number of ICU stays | Up to approximately 6 years
  Described as the cumulative number of days during ICU stays.
ICU days | Up to approximately 6 years
Number of patients with OP visit | Up to approximately 6 years
  OP services include office visits, skilled-nursing facility, home care, durable medical equipment, and other services that are not included in IP stays or ER visits.
Number of OP visits | Up to approximately 6 years
Number of patients with ER visit | Up to approximately 6 years
Number of ER visits | Up to approximately 6 years
Healthcare reimbursement costs | Up to approximately 6 years
  Healthcare reimbursement costs were defined as the amount paid by Medicare to the provider for medical services.
Overall survival (OS) | Up to approximately 6 years
  OS was defined as the time from administration of CAR-T therapy to death due to any cause.
Time to next treatment (TTNT) or death | Up to approximately 6 years
  TTNT was defined as the time from administration of CAR-T therapy to the initiation of the next line of treatment or death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, East Hanover, New Jersey, United States